CLINICAL TRIAL: NCT04292288
Title: Hypercalcemia After Paraffin Oil Injection: Aetiology, Pathogenesis and Possible Treatment Options
Brief Title: Hypercalcemia After Paraffin Oil Injection
Status: Recruiting | Type: Observational
Sponsor: Martin Blomberg Jensen (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, Group leader, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-19010297
Record Dates: First submitted 2019-09-26; First posted 2020-03-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Hypercalcemia; Granuloma
MeSH Terms: conditions — Hypercalcemia; Granuloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Foreign body granuloma: men injecting paraffin oil
  Interventions: Diagnostic Test: Biochemical observational

INTERVENTIONS:
Diagnostic Test: Biochemical observational — no intervention - observational

SUMMARY:
Today, there is an increased use of non-medical, invasive cosmetic treatments globally without sufficient awareness of possible health risks. A particular problem is young men injecting large amounts of paraffin oil into skeletal muscles especially on upper arms and chest to increase the visible size of the muscles. Several case reports have suggested that intramuscular injection of paraffin oil induces foreign body reaction and granuloma formation and subsequently hypercalcemia. Our hypothesis is that increased generation of activated vitamin D (1,25(OH)2D3) in the marcrophages may be responsible for the persistent hypercalcemia. Now trhe investigators want to include a large group of men who injected 100-10.000 ml paraffin oil to identify risk factors for developing hypercalcemia and try to understand the pathogenesis of the disease. Additionally, granuloma tissue from selected patients will be cultured ex vivo to investigate whether they produce 1,25(OH)2D3 or PTHrP and to test which drugs can most effectively be used to lower calcium levels in these men. Subsequently, we will try to stratify the men according to the severity of the changes in calcium homeostasis as we suggest that this stratification will be the basis for future intervention trials

DETAILED DESCRIPTION:
Today, there is an increased use of non-medical, invasive cosmetic treatments globally without sufficient awareness of possible health risks. A particular problem is young men injecting large amounts of paraffin oil into skeletal muscles especially on upper arms and chest to increase the visible size of the muscles. Several case reports have suggested that intramuscular injection of paraffin oil induces foreign body reaction and granuloma formation. The formation of granuloma probably precedes the marked hypercalcemia that often develops and appears to be difficult to treat. The largest study to date included 14 men and showed that practically all men developed serious hypercalcemia, but the etiology was unclear. Foreign body granulomas are like other granulomatous diseases such as Tuberculosis or sarcoidosis rich in macrophages, (ref) and it has been proposed that increased generation of activated vitamin D (1,25(OH)2D3) in the marcrophages may be responsible for the persistent hypercalcemia.

Calcium homeostasis is tightly regulated primarily by vitamin D, Parathyroid hormone (PTH) and Fibroblast growth factor 23 (FGF23) that rapidly modifies intestinal absorption, renal excretion and calcium mobilization from the skeletal compartment in response to immediate changes in serum calcium (ref). Vitamin D (cholecalciferol) is normally formed by UV-B radiation of the skin and requires two enzymatic reactions before it can bind and activate the vitamin D receptor (VDR). Conversion of cholecalciferol to 25-hydroxydvitamin (25OHD) is the first activation step; it is un-regulated and generally exerted by the hepatic CYP2R1. 25OHD is not biologically active and must undergo 1-alpha hydroxylation by renal CYP27B1 to form the active metabolite 1,25(OH)2D3. The main actions of 1,25(OH)2D3 is to promote calcium and phosphate absorption and decrease calcium excretion until inactivated by CYP24A1. 1,25(OH)2D3 is also a powerful inhibitor of PTH and inducer of FGF23, which ensures an important feedback-loop to maintain an adequate vitamin D status (ref). PTH which is a potent inducer of CYP27B1, mobilizes calcium and phosphate from the skeleton and increases phosphate excretion. In contrast, FGF23 that inhibits CYP27B1, induces the in-activating CYP24A1 and promotes phosphate excretion. Almost all organs has the ability to activate, respond to, and inactivate vitamin D because CYP27B1, VDR and CYP24A1 are expressed also in most non-renal tissues. However, regulation of CYP27B1 and CYP24A1 is strikingly different in these organs where high intracellular levels of 1,25(OH)2D3 activates VDR that induces transcription of CYP24A1 and thereby increases in-activation to restore normal intracellular levels of all vitamin D metabolites. This autoregulatory control of vitamin D metabolites secures under normal circumstances that high concentrations of 1,25(OH)2D3 are not released into circulation. Regulation of vitamin D homeostasis is different in the macrophages present in granulomas because they retain a splice variant of CYP24A1 that is not upregulated in response to high 1,25(OH)2D3 levels, which in part explains the increased release of 1,25(OH)2D3 in granulomatosis disease. Another important issue is aberrant regulation of CYP27B1 in macrophages, which is induced by inflammatory signals such as interleukin-2 and TNF-alpha rather than PTH. Previous case reports have detected CYP27B1 expression in granuloma tissue by immunohistochemistry. However, these findings have to our knowledge never been corroborated by a more comprehensive analysis of enzyme activity and a recent study questioned the etiology because most men with granulomas had normal levels of 1,25(OH)2D3 in serum (ref).

In the present study the investigators want to include a large group of men who injected 100-10.000 ml paraffin oil to identify risk factors for developing hypercalcemia and try to understand the pathogenesis of the disease. Additionally, granuloma tissue from selected patients will be cultured ex vivo to investigate whether they produce 1,25(OH)2D3 or PTHrP and to test which drugs can most effectively be used to lower calcium levels in these men. Subsequently, elucidate whether it is possible to stratify the men according to the severity of the changes in calcium homeostasis as such a stratification may be required prior to and form the basis for future intervention trials

ELIGIBILITY:
Inclusion Criteria: - previous injection of paraffin oil into the body

-

Exclusion Criteria: - inability to walk

* inability to understand the consequences of inclusion
* incurable cancer disease

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — no females
Study Population: Up to 200 people (predominantly men) <80 years will be included. Inclusion takes place at Endocrinological Section, Medical Department O, Herlev Hospital in connection with an outpatient visit. After initial discussions, reflection time and acceptance of participation in the study, extended blood tests are taken in connection with the pre-planned outpatient visits.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Hypercalcemia | determined 2-10 years after paraffin oil injection (first visit)
  the number of men with elevated ionized calcium (above 1.32 mmol/l)
production of 1,25OHD3 | ex vivo culture experiments of human granuloma tissue for 48 to 72 hours
  production of 1,25OHD3 determined in media from granuloma tissue culture compared with kidney culture by ELISA platform

SECONDARY OUTCOMES:
hypercalciuria | determined 2-10 years after paraffin oil injection
  calcium excretion determined by spot or 24 hour urine
change in serum 1,25OH2D3 | determined 2-10 years after paraffin oil injection (first visit)
  differences in calcitriol production or conversion rate 1,25OH2D3/25OHD that reflects how active the enzyme is
nephrolithiasis | determined 2-10 years after paraffin oil injection (first visit)
  obtained by interview -anamnesis and preferably supported by jorunal of CT report on nephrolithiasis
Overall change in calcium homeostasis | determined 2-10 years after paraffin oil injection (first visit)
  changes in calcium, PTH, alkaline phosphatase and 1,25OHD depending on oil injected, varm/cold
inflammatory response | determined 2-10 years after paraffin oil injection (first visit)
  changes in inflammatory markers IL2R, ferritin, ACE
Bone formation and resorption | determined 2-10 years after paraffin oil injection (first visit)
  Serum levels of alkaline phosphatase, C-terminal telopeptide of type I collagen (CTX-I) and N-terminal propeptide of type I procollagen (PINP)
renal function | determined 2-10 years after paraffin oil injection (first visit)
  change in GFR, creatinine, Urea
calciphylaxis | determined 2-10 years after paraffin oil injection (first visit)
  risk determined by Calcium - phosphate product
Suppressed PTH | determined 2-10 years after paraffin oil injection (first visit)
  PTH lower than lower reference (2)
suppression of 1,25OHD3 production | ex vivo culture experiments of human granuloma tissue exposed to treatments for 48 and 72 hours
  production of 1,25OHD3 released into the media from granuloma culture suppressed by different treatments in vitro
production of PTHrP | ex vivo culture experiments of human granuloma tissue for 48 and 72 hours
  PTHrP production in granuloma determined by ELISA platform

CONTACTS AND LOCATIONS:
Overall Officials: Ebbe Eldrup, Study Chair — Herlev
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No